CLINICAL TRIAL: NCT00188799
Title: A Clinical Study of X-ray Volume Imaging to Evaluate the Daily Set-up Accuracy of Conformal Prostate Radiotherapy
Brief Title: Xray Volume Imaging (Cone Beam CT) - Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Canadian Association of Radiation Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0483-CE; Abbott-CARO Uro-OncologicAward
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: daily Xray volume imaging for planning radiotherapy

SUMMARY:
Conformal dose escalated radiotherapy was adopted as the standard treatment technique at PMH for intermediate risk patients with localised disease in 1997. This technique provides a much smaller margin of error for treatment set-up and delivery than with conventional techniques. One way to ensure the accuracy of treatment delivery is to image the prostate position daily, prior to therapy, to allow for appropriate set-up corrections. To do so, imaging markers are implanted into the prostate under guided ultrasound (a standard procedure at PMH). However, there are disadvantages in using imaging markers which include added time to the treatment planning process, and an invasive procedure with a potential for discomfort, bleeding and infection. This study will investigate and compare X-ray volume imaging to the gold standard imaging markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate
* Patient undergoing escalated dose conformal external beam radiotherapy.
* Patient has low or intermediate risk prognostic factors: all of PSA <21, Gleason score <8, clinical T category <T3, clinical N category 0 or X, M category 0 or X.
* Informed consent

Exclusion Criteria:

* No diagnosis of adenocarcinoma of the prostate
* Patient not undergoing escalated dose conformal radiotherapy
* Patient does not have low or intermediate risk prognostic factors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-11; Study Completion 2004-11

PRIMARY OUTCOMES:
To evaluate he feasibility of daily X-ray volume imaging during conformal radiotherapy.

SECONDARY OUTCOMES:
To provide preliminary data concerning the relative utility of daily X-ray volume image matching compared to fiducial marker image matching.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Catton, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada